CLINICAL TRIAL: NCT06356233
Title: Phenotyping and Identification of Biological Markers in STXBP1 Encephalopathy
Acronym: FIMBEX
Status: Not yet recruiting | Type: Observational
Sponsor: Fundación Iniciativa para las Neurociencias (FINCE) (Other)
Responsible Party: Principal Investigator, Adrián Valls Carbó, MD, Fundación Iniciativa para las Neurociencias (FINCE)
Other Study IDs: FIMBEX
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: STXBP1 Encephalopathy With Epilepsy
Keywords: STXBP1
MeSH Terms: conditions — Epileptic Encephalopathy, Early Infantile, 4

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention will be performed — No intervention will be performed

SUMMARY:
This is a prospective observational study to evaluate the phenotype of 10 patients under 10 years of age with developmental epileptic encephalopathy due to mutation of the STXBP1 gene. The study will consist of a clinical and neurodevelopmental evaluation, magnetic resonance imaging, prolonged electroencephalogram, cardiological study, and analysis of biomarkers in cerebrospinal fluid. These patients will be followed up for 3 years. The aim of the study is, knowing the baseline phenotype, to analyse the response to commonly used drugs and to anticipate the response to different drugs available on the market in this group of patients based on clinical and biomarker assessment (EEG, MRI and study of specific proteins and neurotransmitters in plasma, urine and CSF).

ELIGIBILITY:
Inclusion Criteria:

* Patients under 10 years of age with confirmed mutation for STXBP1. In cases where the diagnostic technique for the mutation is not optimal, a trio exome will be performed to confirm the mutation.

Exclusion Criteria:

* Presence of functional disability that prevents the neuropsychological study from being carried out and absence of a reliable informant for the patient.

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients under 10 years of age with confirmed mutation for STXBP1 willing to collaborate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
CSF biomarkers | Baseline, 1 year and 2 years
EEG markers | Baseline, 1 year and 2 years
MRI markers | Baseline, 1 year and 2 years

SECONDARY OUTCOMES:
Clinical phenotype | Baseline, 1 year and 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ruber Internacional, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No